CLINICAL TRIAL: NCT05449106
Title: Evaluation of Clinical Outcomes of Unruptured Brain Arteriovenous Malformations Treated With Medical Management Alone Based on Multimodal Computer Tomography: A Long-term Multicenter Prospective Cohort Study
Brief Title: Evaluation of Clinical Outcomes of Unruptured bAVMs Treated With Medical Management Alone Based on Multimodal CT
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Hospital (Other Government); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Other Study IDs: KY2022-054-02
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Brain Arteriovenous Malformations
Keywords: Unruptured arteriovenous malformations; Multimodal CT; Machine learning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate the role of multimodal CT in evaluating and predicting different clinical outcomes in patients with unruptured brain arteriovenous malformations with medical management alone.

This study will be undertaken in the following aspects:

1. Morphological, structural and imaging histological signal analysis based on multimodal CT to explore the relationship between imaging features and different clinical outcomes of bAVMs.
2. Hemodynamic and flow pattern analysis of local and peripheral bAVMs based on multimodal CT to explore the association between blood flow features and different clinical outcomes.
3. Based on multimodal CT and deep learning algorithms to create an automated segmentation model for bAVMs and a prediction model for distinct clinical outcomes.

The obtained patient information includes: Baseline information, CT, MRI, DSA (Optional), and follow-up information. Follow-up will be undertaken at 6 months, 12 months, 24 months and 36 months after enrollment with the following primary observation.

Main observation endpoints:

1. Hemorrhage events associated with bAVMs
2. New epilepsy symptoms or exacerbations
3. New neurological dysfunction(including motor dysfunction, cognitive dysfunction, etc).

DETAILED DESCRIPTION:
This study is a Long-term, multi-center, prospective registry study, and was supported by China National Key Research and Development Program Project No. 2021YFC2500502.

The purpose of this study is to investigate the role of multimodal Computer Tomography(CT) in evaluating and predicting different clinical outcomes in patients with unruptured brain arteriovenous malformations with medical management alone.

This study will be undertaken in the following aspects:

1. Morphological, structural and imaging histological signal analysis based on multimodal CT to study the relationship between imaging features and different clinical outcomes of bAVMs.
2. Hemodynamic and flow pattern analysis of local and peripheral bAVMs based on multimodal CT to explore the association between blood flow features and different clinical outcomes.
3. Based on multimodal CT and deep learning algorithms to create an automated segmentation model for bAVMs and a prediction model for distinct clinical outcomes.
4. To compare the efficacy of multimodal CT and MRI in evaluating the clinical outcomes of unruptured cerebral arteriovenous malformations.

The obtained patient information includes:

1. Baseline information
2. CT images: including non-contrast CT(NCCT), CT Angiography, CT perfusion
3. Magnetic Resonance Imaging(MRI): including T1-weighted image, T2-weighted image, T2-FLAIR, Time of Flight MR angiography(TOF-MRA), diffusion-weighted imaging(DWI), susceptibility weighted imaging(SWI)
4. Digital subtraction angiography(DSA, optional)
5. Follow-up information: follow-up will be undertaken at 6 months, 12 months, 24 months and 36 months after enrollment with the following primary observation.

Main observation endpoints:

1. Hemorrhage events associated with bAVMs, ensuring by CT scan;
2. New epilepsy symptoms or exacerbations, ensuring by consultation or EEG ;
3. New neurological dysfunction(including motor dysfunction, cognitive dysfunction, etc), ensuring by consultation, physical examination or any radiology examination.

Inclusion criteria

1. Patients with confirmed diagnosis of bAVMs in the cerebrum, basal ganglia, thalamus, corpus callosum, cerebellum and brainstem;
2. Patients with no history of previous bAVM related hemorrhage confirmed by CT examination, or have radiographic examination completed prior to the hemorrhage.
3. Patients with radiographic examinations before any treatment;

Exclusion criteria.

1. Patients with simple arteriovenous fistula;
2. Patients with combined dural arteriovenous fistula;
3. Arteriovenous malformations occurring in the spinal cord;
4. Pregnant patients were not included in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed diagnosis of brain arteriovenous malformations in the brain, basal ganglia, thalamus, corpus callosum, cerebellum and other locations.
2. Patients with no history of previous arteriovenous malformation-related hemorrhage and no arteriovenous malformation-related hemorrhage confirmed by CT examination.
3. Patients with Radiographic examinations completed without any treatment

Exclusion Criteria:

1. Patients with simple arteriovenous fistula.
2. Patients with combined dural arteriovenous fistulas.
3. Arteriovenous malformations occurring in the spinal cord.
4. Pregnant patients were not included in this study.

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with the diagnosis of AVM was confirmed with Digital Subtraction Angiography (DSA) , Magnetic Resonance Imaging(MRI), or Computed Tomography Angiography, eligible for enrollment criteria and have images that were acquired without any intervention.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2027-05-25 (Estimated); Study Completion 2032-05-25 (Estimated)

PRIMARY OUTCOMES:
Number of participants with rupture events | 3 years after enrollment
  Arteriovenous malformation rupture during follow-up before treatment
Number of participants with epilepsy Progression | 3 years after enrollment
  Progression of seizure symptoms during follow-up, including but not limited to more frequent seizures, worsening of symptoms, etc.
Number of participants with new onset neurological dysfunction | 3 years after enrollment
  New neurological deficits during the follow-up period, including motor deficits, cognitive deficits, etc.

SECONDARY OUTCOMES:
Number of participants receiving treatment | 3 years after enrollment
  Patients receiving any form of intervention during the follow-up period will stop the follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Dong Zhang, Doctor, Study Chair — Beijing Tiantan Hospital, Beijing Hospital; Shaosen Zhang, Doctor, Study Director — Beijing Tiantan Hospital; Guosheng Zhou, Principal Investigator — The First Affiliated Hospital of Zhengzhou University; Yongbo Yang, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (4):
- China (4):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu